CLINICAL TRIAL: NCT06454032
Title: Effect of 12-week Fitness Walking Programme on Sex Hormone Levels and Risk Factors for Metabolic Syndrome in Postmenopausal Women
Brief Title: Effect of 12-week FW Programme on Sex Hormone Levels and Risk Factors for MS in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EOFWOSHLARFMSIPP
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Postmenopause Women
Keywords: Exercise; Postmenopause; Women's health; Metabolism; Sex hormone
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fitness walking group (Experimental)
  Interventions: Behavioral: Fitness walking
- Control group (Sham Comparator)
  Interventions: Behavioral: Maintained lifestyle

INTERVENTIONS:
Behavioral: Fitness walking — Fitness walking for 12 weeks.
  Arms: Fitness walking group
Behavioral: Maintained lifestyle — Maintained their normal lifestyle, without exercise intervention.
  Arms: Control group

SUMMARY:
Postmenopausal women were separated into two groups: one participating in a 12-week fitness walking programe as the fitness walking group, and the other maintaining their regular lifestyle as the control group. The study evaluated alterations in health markers and examined the correlation between metabolic syndrome risk factors and sex hormone levels before and after the intervention.

DETAILED DESCRIPTION:
According to the inclusion and exclusion criteria, our study invlved postmenopausal women aged from 50 to 69 years old. After the selection process, baseline assessments were conducted, including evaluations of metabolic syndrome risk factors, body morphology measurements, sex hormone levels, and cardiopulmonary exercise testing. Participants were then randomly assigned to either the fitness walking group or the control group using a random number table. Participants in the fitness walking group completed a 12-week fitness walking program, while those in the control group maintained their usual lifestyle without any intervention. During the post-intervention assessment, all baseline measurements were repeated to evaluate changes in the previously measured indicators.

ELIGIBILITY:
Inclusion Criteria:

* (1) Participants were entirely voluntary and capable of completing the full 12-week intervention process.
* (2) Participants were postmenopausal women aged between 50 and 69 years.
* (3) Participants had been postmenopausal for over 12 months and had not received exogenous estrogen supplementation post-menopause.

Exclusion Criteria:

* (1) Participants had a history of acute or chronic musculoskeletal disorders, cardiovascular diseases, diabetes, or other conditions that might impact their ability to engage in the intervention.
* (2) Participants had recent hormone treatment, anti-inflammatory medication use, or other medications affecting blood indices.
* (3) Participants experienced unstable body weight (fluctuations exceeding 2.5 kg) in the past three months.
* (4) Participants were concurrently enrolled in other intervention studies or maintained regular exercise routines.
* (5) Participants had smoking or alcohol consumption habits.

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-16 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure (SBP) | At the beginning-at 12 weeks.
  The change of SBP before and after intervention
Diastolic blood pressure (DBP) | At the beginning-at 12 weeks.
  The change of DBP before and after intervention
Waist circumference (WC) | At the beginning-at 12 weeks.
  The change of WC before and after intervention
Fasting blood glucose (FBG) | At the beginning-at 12 weeks.
  The change of FBG before and after intervention
Triglycerides (TG) | At the beginning-at 12 weeks.
  The change of TG before and after intervention
High-density lipoprotein cholesterol (HDL-C) | At the beginning-at 12 weeks.
  The change of HDL-C before and after intervention

SECONDARY OUTCOMES:
Oestradiol (E2) | At the beginning-at 12 weeks.
  The change of E2 before and after intervention
Testosterone (T) | At the beginning-at 12 weeks.
  The change of T before and after intervention
Sex hormone-binding globulin (SHBG) | At the beginning-at 12 weeks.
  The change of SHBG before and after intervention
Dehydroepiandrosterone sulphate (DHEA-S) | At the beginning-at 12 weeks.
  The change of DHEA-S before and after intervention
Maximal oxygen uptake (VO2max) | At the beginning-at 12 weeks.
  The change of VO2max before and after intervention
Body weight (BW) | At the beginning-at 12 weeks.
  The change of BW before and after intervention
Height | At the beginning-at 12 weeks.
  The change of height before and after intervention
Body mass index (BMI) | At the beginning-at 12 weeks.
  The change of BMI before and after intervention

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - School of Sports Medicine and Rehabilitation, Beijing Sport University, Beijing
  - School of Sports Medicine and Rehabilitation, Beijing